CLINICAL TRIAL: NCT04776187
Title: Safety Evaluation of Linear and Macrocyclic Gadolinium-Based Contrast Agents for Patients With Mild to Moderate Renal Insufficiency Undergoing Enhanced Magnetic Resonance Imaging (Interventional Prospective Study) Clinical Trial Protocol
Brief Title: Safety Evaluation of Linear and Macrocyclic Gadolinium Based Contrast Agents for Patients With Mild to Moderate Renal Insufficiency Undergoing Enhanced Magnetic Resonance Imaging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gadolinium 1.0
Record Dates: First submitted 2021-01-11; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Nephrogenic Fibrosing Dermopathy
Keywords: Humans; gadodiamide; MRI; Renal Insufficiency; Drug-Related Adverse Reactions
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy; Renal Insufficiency | interventions — gadodiamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gadodiamide (Active Comparator): Patients who have undergone contrast-enhanced MRI using Gadodiamide contrast agent for clinical purposes.
  Generic name: Gadodiamide Injection; Product name: OMNISCAN; Sample specifications: 15ml: 4.305g (a sterile solution containing 287mg/ml gadodiamide).
  Interventions: Drug: Gadodiamide
- Gadoteric Acid Meglumine Salt (Experimental): Patients who have undergone contrast-enhanced MRI using Gadoteric Acid Meglumine Salt contrast agent for clinical purposes.
  Generic name: Gadoteric Acid Meglumine Salt Injection; Commodity name: Jia Di Xian; Sample specifications: 15ml: 5.654g (a sterile solution containing 377mg/ml gadoteric acid meglumine salt).
  Interventions: Drug: Gadoteric Acid Meglumine Salt

INTERVENTIONS:
Drug: Gadodiamide — Gadodiamide Injection(OMNISCAN™)
  Arms: Gadodiamide
Drug: Gadoteric Acid Meglumine Salt — Gadoteric Acid Meglumine Salt Injection(Jia Di Xian™)
  Arms: Gadoteric Acid Meglumine Salt

SUMMARY:
The purpose of this study is to evaluate the safety of linear and macrocyclic gadolinium-based contrast agents for patients with mild to moderate renal insufficiency. The study will compare the incidence of adverse events of gadodiamide and gadoteric Acid Meglumine Salt for patients with mild to moderate renal insufficiency undergoing enhanced magnetic resonance imaging.

DETAILED DESCRIPTION:
According to the requirements of the study, 600 cases of patients with mild to moderate renal insufficiency were enrolled. Gadodiamide and Gadoteric acid meglumine salt were used for enhanced MRI. Observe the adverse reactions within 60 minutes of using the gadolinium contrast agents; follow up by telephone at 3, 6, 12, and 24 months after the inspection. The primary endpoint is the incidence of the various adverse events, and the secondary endpoints are changes of serum creatinine and inflammatory factors (TNF-α, hs-CRP, IL-6) before and after CE-MRI, patient skin examination and evaluation (evaluation of relevant indicators of skin biopsy).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old who require gadolinium-based CE-MRI;
2. Patients with renal function 30ml/min/1.73m2≤eGFR<90/min/1.73m2;
3. Patients who are able and willing to comply with the required inspection requirements.

Exclusion Criteria:

1. Patient who experienced allergic reactions to previous gadolinium-based contrast agents;
2. Patient who had used gadolinium-based contrast agents within 3 months;
3. Patient with acute renal failure;
4. Patient who cannot comply with or cannot tolerate the necessary fluid replenishment procedures;
5. Patient with major mental illness, impaired consciousness, or other diseases considered by researchers to affect observation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of various adverse events | From the date of contrast injection to the incidence of adverse events, assessd up to 60 minutes
The incidence of various adverse events | From the date of contrast injection to the incidence of adverse events, assessd up to 3 months
The incidence of various adverse events | From the date of contrast injection to the incidence of adverse events, assessd up to 6 months
The incidence of various adverse events | From the date of contrast injection to the incidence of adverse events, assessd up to 12 months
The incidence of various adverse events | From the date of contrast injection to the incidence of adverse events, assessd up to 24 months

SECONDARY OUTCOMES:
Changes of serum creatinine before and after CE-MRI at 3 days | From the date of contrast injection to the changes of serum creatinine before and after CE-MRI, assessed up to 3 days
Changes of TNF-α before and after CE-MRI at 3 days | From the date of contrast injection to the changes of TNF-α before and after CE-MRI, assessed up to 3 days
Changes of hs-CRP before and after CE-MRI at 3 days | From the date of contrast injection to the changes of hs-CRP before and after CE-MRI, assessed up to 3 days
Changes of IL-6 before and after CE-MRI at 3 days | From the date of contrast injection to the changes of IL-6 before and after CE-MRI, assessed up to 3 days
Evaluation of relevant indicators of skin biopsy | From the date of contrast injection to the clinical manifestations appear, assessed up to 24 months
  proliferation of fibroblasts in subcutaneous tissue, thickening of collagen fiber bundles

CONTACTS AND LOCATIONS:
Locations (1):
- Lishui Central Hospital, Lishui, Zhejiang, China

DOCUMENTS (2):
  • Informed Consent Form (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT04776187/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT04776187/Prot_SAP_001.pdf